CLINICAL TRIAL: NCT00584532
Title: Effects of a Genistein Concentrated Polysaccharide (GCP) on Patients With a Diagnosis of Prostate Cancer on Active Surveillance.
Brief Title: Effects of a Genistein Concentrated Polysaccharide (GCP) for Prostate Cancer on Active Surveillance.
Acronym: GCP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Robert Hackman, PhD, University of California, Davis - Department of Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 281609
Record Dates: First submitted 2007-12-22; First posted 2008-01-02 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2007-12

CONDITIONS: Prostate Cancer
Keywords: Localized; Prostate; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — genistein combined polysaccharide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): A=Placebo ARM of Study
  Interventions: Drug: Placebo
- B (Active Comparator): B=GCP Capsules. Ten 500 mg capsules per day for a total of 5 grams a day.
  Interventions: Drug: GCP - Genistein Combined Polysaccharide

INTERVENTIONS:
Drug: Placebo — 10 Placebo Capsules taken orally every day.
  Other Names: Placebo capsules (contain cellulose only)
  Arms: A
Drug: GCP - Genistein Combined Polysaccharide — Ten 500 mg capsules given orally per day. Total of 5 grams per day per patient.
  Arms: B

SUMMARY:
Genistein Combined Polysaccharide (GCP) may play a role as a secondary chemopreventive agent in the treatment of localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be male and have a pathological diagnosis of prostate cancer
* Pathological diagnosis of prostate cancer must be confirmed and on file with CRA prior to study entry.
* No treatment (surgery, radiation, or hormones) prior to study entry.
* PSA between 2.0 and 10.0 ng/ml.
* If PSA is >10.0, patient must have been on Active Surveillance for 12 months prior to study initiation.
* No known allergy to soy or soy products.
* The patient is not currently taking more than 2 grams of genistein a day in nutritional or diet enhancing supplements (OTC supplements).
* Participant has not been on any previous GCP clinical trial.
* Normal Chemistry values prior to study entry.

Exclusion Criteria:

* No pathological documentation of prostate cancer.
* Prior treatment for prostate cancer.
* PSA >10.0 ng/ml but not on Active Surveillance for 12 months.
* Allergy to soy or soy products.
* Abnormal chemistry values.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-11; Primary Completion 2005-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Decrease in PSA levels in men on GCP | 6 Months

SECONDARY OUTCOMES:
Increased PSA Doubling Time (PSADT)in men on GCP. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hackman, MD, Principal Investigator — University of California, Davis - Dept. of Nutrition